CLINICAL TRIAL: NCT03433105
Title: To Investigate the Prognostic Value of Oxygen Uptake in Weaning of Patients From Prolonged Mechanical Ventilation
Brief Title: Oxygen Uptake in Weaning of Patients From Prolonged Mechanical Ventilation
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201710003RINB
Record Dates: First submitted 2018-01-23; First posted 2018-02-14 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2019-09

CONDITIONS: Ventilator Weaning
Keywords: oxygen uptake; prolonged mechanical ventilation; weaning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1/patients with tracheostomy tubes and prolonged MV use: Patients who have tracheostomy tubes and with prolonged mechanical ventilation

SUMMARY:
1.Research hypothesis: during weaning patient from prolonged mechanical ventilation, if the work load caused by weaning was below the patient's AT, oxygen uptake will be constant. Otherwise, if the work load was above the patient's AT, the oxygen uptake will increase.

1. Patient: who have tracheostomy tubes and with prolonged mechanical ventilation
2. Measurement: oxygen uptake(V̇O2) and respiratory mechanics during the spontaneous breathing trials
3. Outcome: Correlation between the oxygen uptake(V̇O2) and the weaning outcome

2.Specific aims:

1. to investigate the prognostic value of oxygen uptake in weaning patients from prolonged mechanical ventilation
2. Subgroup analysis may suggest which weaning protocol potentially benefit the most for each population group (cardiovascular disease, chronic pulmonary disease, neuromuscular disease, cerebrovascular disease)

ELIGIBILITY:
1. Inclusion criteria:

   Adult >20 y/o Total duration of mechanical ventilation ≥ 10 days Received tracheostomy Defervescence Meeting the criteria of weaning phase (see supplementary protocols)
2. Exclusion criteria FiO2 >50 % Unstable hemodynamics Fever with active infection No spontaneous respiratory drive Dynamic airway collapse

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who have tracheostomy tubes and with prolonged mechanical ventilation
Sampling Method: Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2020-08-14 (Actual); Study Completion 2020-08-14 (Actual)

PRIMARY OUTCOMES:
Measurement of oxygen uptake (V̇O2) | up to 12 hours during the spontaneous breathing trial
  oxygen uptake during the spontaneous breathing trial

CONTACTS AND LOCATIONS:
Overall Officials: Yao-Wen Kuo, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan